CLINICAL TRIAL: NCT01147900
Title: Evaluation of GSK Biologicals' Boostrix™ in Healthy Adults, 10 Years After Previous Booster Vaccination
Brief Title: Evaluation of Boostrix™10 Years After Previous Booster Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113055
Record Dates: First submitted 2010-05-20; First posted 2010-06-22 (Estimated); Results first posted 2013-10-08 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2016-09

CONDITIONS: Acellular Pertussis; Tetanus; Diphtheria
Keywords: Immune persistence; Boostrix; dTpa booster study
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — Boostrix

ARMS (3):
- Boostrix-REF Group (Experimental): Subjects in this group were healthy adult subjects aged 18 to 28 years at the time of enrolment and with previous completed primary and booster vaccination with a diphtheria-tetanus-whole cell pertussis vaccine completed by one additional booster dose of Boostrix™ vaccine, reference formulation, at Day 0 in GSK 263855/029 study. These subjects received, as part of this NCT01147900 study, one further booster dose of Boostrix™ vaccine, reference formulation, at Year 10, 10 years after booster vaccination in the GSK 263855/029 study. The Boostrix™ vaccine was administered intramuscularly in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Boostrix™
- Boostrix-US Group (Experimental): Subjects in this group were healthy adult subjects aged 18 to 28 years at the time of enrolment and with previous completed primary and booster vaccination with a diphtheria-tetanus-whole cell pertussis vaccine completed by one additional booster dose of Boostrix™ vaccine, United States(US)-marketed formulation, at Day 0 in GSK 263855/029 study. These subjects received, as part of this NCT01147900 study, one further booster dose of Boostrix™ vaccine, US-marketed formulation, at Year 10, 10 years after booster vaccination in the GSK 263855/029 study. The Boostrix™ vaccine was administered intramuscularly in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Boostrix™-US formulation
- Boostrix-INV Group (Experimental): Subjects in this group were healthy adult subjects aged 18 to 28 years at the time of enrolment and with previous completed primary and booster vaccination with a diphtheria-tetanus-whole cell pertussis vaccine completed by one additional booster dose of Boostrix™ vaccine, investigational formulation, at Day 0 in GSK 263855/029 study. These subjects received, as part of this NCT01147900 study, one further booster dose of Boostrix™ vaccine, reference formulation, at Year 10, 10 years after booster vaccination in the GSK 263855/029 study. The Boostrix™ vaccine was administered intramuscularly in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Boostrix™

INTERVENTIONS:
Biological: Boostrix™ — Intramuscular, single dose
  Arms: Boostrix-INV Group; Boostrix-REF Group
Biological: Boostrix™-US formulation — Intramuscular, single dose
  Arms: Boostrix-US Group

SUMMARY:
The purpose of the study is to evaluate the immunogenicity, safety and reactogenicity of a dTpa (Boostrix™ vaccine) booster dose given 10 years after the previous vaccination with dTpa in GSK 263855/029 study. Only subjects who were part of the primary study will be invited to participate in this study.This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate study (see reference).

DETAILED DESCRIPTION:
All subjects will receive a booster dose of the vaccine that they received in their primary study. Subjects who received the investigational vaccine formulation, will receive Boostrix™ in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Male or female subjects who have received Boostrix™, Boostrix™-US formulation or the investigational vaccine formulation in the study 263855/029.
* Written informed consent obtained from the subject. Additional criteria to be checked before the booster vaccination.
* Healthy subjects as established by medical history and clinical examination.
* Female subjects of non-childbearing potential may receive the booster vaccine.
* Female subjects of childbearing potential may receive the booster vaccine, if the subject:

  * practices/has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * agrees to continue adequate contraception during the entire booster epoch.

Exclusion Criteria:

Exclusion criteria to be checked at study entry:

* Previous booster vaccination against diphtheria, tetanus, or pertussis since the dose received in the study 263855/029.
* History of diphtheria, tetanus, or laboratory confirmed pertussis disease.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Occurrence of transient thrombocytopenia or neurological complications following an earlier immunisation against diphtheria and/or tetanus.
* Occurrence of any of the following adverse event after a previous administration of a DTP vaccine :

  * hypersensitivity reaction to any component of the vaccine,
  * encephalopathy of unknown aetiology occurring within seven days following previous vaccination with pertussis-containing vaccine,
  * fever >= 40 °C (axillary temperature) within 48 hours of vaccination not due to another identifiable cause,
  * collapse or shock-like state within 48 hours of vaccination,
  * convulsions with or without fever, occurring within three days of vaccination.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.

Additional exclusion criteria to be checked for subjects before the booster vaccination administration:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to booster vaccination, or planned administration during the active study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster dose or planned administration during the study period.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C on oral, axillary or tympanic setting.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2010-06-15; Primary Completion 2012-05-08 (Actual); Study Completion 2012-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Wilrijk

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Vandermeulen C, Theeten H, Rathi N, Kuriyakose S, Han HH, Sokal E, Hoppenbrouwers K, Van Damme P. Decennial administration in young adults of a reduced-antigen content diphtheria, tetanus, acellular pertussis vaccine containing two different concentrations of aluminium. Vaccine. 2015 Jun 12;33(26):3026-34. doi: 10.1016/j.vaccine.2014.10.049. Epub 2015 Jan 19. PMID 25613716
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113055 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects consisted of those previously vaccinated & boosted in GSK263855/029 study and contacted for participation in this booster (BST) study. Duration of this study was about 19 months, from Year 8.5 (8.5 years post BST in GSK263855/029 study) to one month post BST in this study (Year 10 [10 years post BST in GSK263855/029 study] + one month).
Pre-assignment Details: At Year 8.5, a total of 180 subjects (out of the 478 planned) were enrolled: 54, 60 and 66 subjects in the Boostrix-REF, Boostrix-US, and Boostrix-INV groups, respectively. At Year 10, a total of 177 subjects (out of the 180 planned) were enrolled: 55, 60 and 62 in the Boostrix-REF, Boostrix-US, and Boostrix-INV groups, respectively.
Period: At Year 8.5
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Started | 54 | 60 | 66
Completed | 54 | 60 | 66
Not Completed | 0 | 0 | 0
Period: At Year 10
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Started | 55 (At Year 10, a total of 177 subjects (out of the 180 planned) were enrolled) | 60 | 62 (At Year 10, a total of 177 subjects (out of the 180 planned) were enrolled.)
Completed | 55 | 59 | 62
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: At Year 8.5, a total of 180 subjects (out of the 478 planned) were enrolled: 54, 60 and 66 subjects in the Boostrix-REF, Boostrix-US, and Boostrix-INV groups, respectively. At Year 10, a total of 177 subjects (out of the 180 planned) were enrolled: 55, 60 and 62 in the Boostrix-REF, Boostrix-US, and Boostrix-INV groups, respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group | Total
Number analyzed (Participants) | 55 | 60 | 66 | 181
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The baseline measure data correspond to Year 8.5.
  Years
    number analyzed (Participants) | 54 | 60 | 66 | 180
    (all) | 22.4 (1.46) | 22.3 (1.20) | 22.3 (1.17) | 22.3 (1.18)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The baseline measure data correspond to Year 10.
  Years
    number analyzed (Participants) | 55 | 60 | 62 | 177
    (all) | 23.5 (1.44) | 23.4 (1.21) | 23.3 (1.17) | 23.4 (1.19)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The baseline measure data correspond to Year 8.5.
  Participants
    number analyzed (Participants) | 54 | 60 | 66 | 180
    Female | 29 | 33 | 39 | 101
    Male | 25 | 27 | 27 | 79
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The baseline measure data correspond to Year 10.
  Participants
    number analyzed (Participants) | 55 | 60 | 62 | 177
    Female | 29 | 31 | 36 | 96
    Male | 26 | 29 | 26 | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Diphtheria and Tetanus
Description: A subject seroprotected against diphtheria/tetanus was defined as a vaccinated subject who had an anti-diphtheria (anti-D)/anti-tetanus (anti-T) antibody concentration greater than or above (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: At Year 8.5
Population: The analysis was performed on the According To Protocol cohort for persistence at Year 8.5, which included all subjects who had received no additional dose of diphtheria, tetanus or pertussis vaccine other than the Boostrix™ booster dose received in the GSK263855/029 study, and for whom serological results were available at Year 8.5.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 59 | 65
Participants
  Anti-D | 53 | 59 | 65
  Anti-T | 54 | 59 | 65

2. Primary Outcome: Concentrations for Anti-D and Anti-T Antibodies.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection cut-off of the assay was 0.1 IU/mL for all antibodies assessed.
Time Frame: At Year 8.5
Population: The analysis was performed on the According To Protocol cohort for persistence at Year 8.5 , which included all subjects who had received no additional dose of diphtheria, tetanus or pertussis vaccine other than the Boostrix™ booster dose received in the GSK263855/029 study, and for whom serological results were available at Year 8.5.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 59 | 65
IU/mL
  Anti-D | 0.912 [0.728 to 1.141] | 1.205 [0.984 to 1.474] | 0.872 [0.711 to 1.068]
  Anti-T | 1.889 [1.585 to 2.251] | 1.991 [1.674 to 2.368] | 1.846 [1.604 to 2.123]

3. Primary Outcome: Number of Seroprotected Subjects Against Diphtheria and Tetanus.
Description: A subject seroprotected against diphtheria/tetanus was defined as a vaccinated subject who had an anti-D/anti-T antibody concentration greater than or above (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: At Year 10
Population: The analysis was performed on the According To Protocol cohort for persistence at Year 10, which included all subjects who had received no additional dose of diphtheria, tetanus or pertussis vaccine other than the Boostrix™ booster dose received in the GSK263855/029 study, and for whom serological results were available at Year 10.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 60 | 61
Participants
  Anti-D | 53 | 60 | 61
  Anti-T | 54 | 60 | 61

4. Primary Outcome: Concentrations for Anti-D and Anti-T Antibodies.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection cut-off of the assay was 0.1 IU/mL.
Time Frame: At Year 10
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 60 | 61
IU/mL
  Anti-D | 0.767 [0.600 to 0.982] | 1.099 [0.882 to 1.370] | 0.681 [0.550 to 0.844]
  Anti-T | 2.008 [1.650 to 2.444] | 2.009 [1.701 to 2.372] | 1.760 [1.518 to 2.041]

5. Primary Outcome: Number of Seropositive Subjects for Anti-pertussis Toxoid (Anti-PT), Anti-pertactin (Anti-PRN) and Anti-filamentous Haemagglutinin (Anti-FHA) Antibodies.
Description: A seropositive subject for anti-PT/anti-PRN/anti-FHA antibodies was defined as a vaccinated subject who had anti-PT/anti-PRN/anti-FHA antibody concentrations greater than or equal to (≥) 5 Enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Year 8.5
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 59 | 65
Participants
  Anti-PT [N=54;59;65] | 42 | 48 | 60
  Anti-FHA [N=54;59;62] | 54 | 59 | 62
  Anti-PRN [N=54;59;65] | 54 | 59 | 65

6. Primary Outcome: Concentrations for Anti-PT, Anti-PRN and Anti-FHA Antibodies.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seropositivity cut-off of the assay was 5 EL.U/mL for all antibodies assessed.
Time Frame: At Year 8.5
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 59 | 65
EL.U/mL
  Anti-PT [N=54;59;65] | 10.933 [7.979 to 14.980] | 13.372 [10.139 to 17.634] | 18.034 [13.812 to 23.545]
  Anti-FHA [N=54;59;62] | 72.653 [57.904 to 91.158] | 96.144 [75.613 to 122.250] | 102.604 [85.687 to 122.861]
  Anti-PRN [N=54;59;65] | 161.349 [121.750 to 213.827] | 179.027 [136.303 to 235.144] | 134.616 [106.266 to 170.528]

7. Primary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN Antibodies.
Description: A seropositive subject for anti-PT/anti-FHA/anti-PRN antibodies was defined as a vaccinated subject who had anti-PT/anti-FHA/anti-PRN antibody concentrations greater than or equal to (≥) 5 Enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Year 10
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 60 | 60
Participants
  Anti-PT [N=52;59;59] | 44 | 49 | 51
  Anti-PRN [N=54;60;60] | 54 | 60 | 60
  Anti-FHA [N=54;60;60] | 54 | 60 | 60

8. Primary Outcome: Concentrations for Anti-PT, Anti-FHA and Anti-PRN Antibodies.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seropositivity cut-off of the assay was 5 EL.U/mL.
Time Frame: At Year 10
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 60 | 60
EL.U/mL
  Anti-PT [N=52;59;59] | 11.627 [8.863 to 15.252] | 13.987 [10.874 to 17.991] | 15.728 [11.760 to 21.034]
  Anti-PRN [N=54;60;60] | 131.814 [98.531 to 176.340] | 158.239 [120.864 to 207.171] | 115.209 [91.288 to 145.398]
  Anti-FHA [N=54;60;60] | 75.574 [61.018 to 93.603] | 98.182 [77.166 to 124.921] | 98.441 [82.710 to 117.165]

9. Primary Outcome: Number of Seroprotected Subjects Against Diphtheria and Tetanus
Description: as for outcome 3
Time Frame: At Year 10 pre booster vaccination (PRE) and at 1 month post Year 10 booster vaccination (POST)
Population: Analysis was done on the According-to-Protocol for immunogenicity at Year 10, which included all evaluable subjects who had received the booster dose of Boostrix™ vaccine, any formulation (at least 9.5 years after the dose administered in GSK263855/029 study) and for whom data concerning immunogenicity outcome measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 59 | 60
Participants
  Anti-D, PRE | 53 | 59 | 60
  Anti-D, POST | 54 | 59 | 60
  Anti-T, PRE | 54 | 59 | 60
  Anti-T, POST | 54 | 59 | 60

10. Primary Outcome: Concentrations for Anti-D and Anti-T Antibodies.
Description: as for outcome 2
Time Frame: At Year 10 pre booster vaccination (PRE) and at 1 month post Year 10 booster vaccination (POST)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 59 | 60
IU/mL
  Anti-D, PRE | 0.767 [0.600 to 0.982] | 1.094 [0.874 to 1.368] | 0.686 [0.552 to 0.853]
  Anti-D, POST | 4.251 [3.646 to 4.957] | 5.226 [4.353 to 6.275] | 4.150 [3.543 to 4.862]
  Anti-T, PRE | 2.008 [1.650 to 2.444] | 1.987 [1.680 to 2.350] | 1.752 [1.508 to 2.037]
  Anti-T, POST | 7.581 [6.523 to 8.809] | 8.456 [7.294 to 9.802] | 8.792 [7.582 to 10.195]

11. Primary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN Antibodies.
Description: A seropositive subject for anti-PT/anti-PRN/anti-FHA antibodies was defined as a vaccinated subject who had anti-PT/anti-PRN/anti-FHA antibody concentrations greater than or equal to (≥) 5 ELISA units per milliliter (EL.U/mL).
Time Frame: At Year 10 pre booster vaccination (PRE) and at 1 month post Year 10 booster vaccination (POST)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 59 | 60
Participants
  Anti-PT, PRE [N=52;58;58] | 44 | 48 | 50
  Anti-PT, POST [N=54;59;60] | 54 | 59 | 60
  Anti-PRN, PRE [N=54;59;59] | 54 | 59 | 59
  Anti-PRN, POST [N=53;59;60] | 53 | 59 | 60
  Anti-FHA, PRE [N=54;59;59] | 54 | 59 | 59
  Anti-FHA, POST [N=53;59;60] | 53 | 59 | 60

12. Primary Outcome: Concentrations for Anti-PT, Anti-FHA and Anti-PRN Antibodies.
Description: as for outcome 8
Time Frame: At Year 10 pre booster vaccination (PRE) and at 1 month post Year 10 booster vaccination (POST)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 59 | 60
EL.U/mL
  Anti-PT, PRE [N=52;58;58] | 11.627 [8.863 to 15.252] | 14.193 [11.003 to 18.306] | 15.650 [11.643 to 21.035]
  Anti-PT, POST [N=54;59;60] | 82.478 [66.951 to 101.606] | 108.094 [87.703 to 133.227] | 123.964 [103.458 to 148.533]
  Anti-PRN, PRE [N=54;59;59] | 131.814 [98.531 to 176.340] | 161.903 [123.574 to 212.120] | 114.226 [90.201 to 144.652]
  Anti-PRN, POST [N=53;59;60] | 445.751 [372.770 to 533.020] | 448.475 [383.748 to 524.120] | 448.839 [379.488 to 530.863]
  Anti-FHA, PRE [N=54;59;59] | 75.574 [61.018 to 93.603] | 96.098 [75.507 to 122.305] | 97.698 [81.891 to 116.555]
  Anti-FHA, POST [N=53;59;60] | 503.532 [426.524 to 594.444] | 592.177 [516.831 to 678.507] | 558.648 [489.266 to 637.869]

13. Primary Outcome: Number of Booster Responders to Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) Antigens.
Description: A booster responder to PT/PRN antigens was defined as either a vaccinated subject seronegative at analysis baseline (Year 10) with anti-PT/anti-PRN antibody concentration greater than or equal to (≥) 5 EL.U/mL at one month post Year 10 booster vaccination, or as a vaccinated subject seropositive at analysis baseline (Year 10) and with anti-PT/anti-PRN antibody concentration with at least a 2-fold increase at one month post Year 10 booster vaccination.
  A seronegative/seropositive subject was defined as a vaccinated subject with anti-PT/anti-PRN antibody concentration ≥/< 5 EL.U/mL.
Time Frame: At 1 month post Year 10 booster vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 46 | 52 | 52
Participants
  Booster responses to anti-PT [N=44;51;51] | 44 | 51 | 48
  Booster responses to anti-PRN [N=45;52;52] | 23 | 29 | 35
  Booster responses to anti-FHA [N=46;52;50] | 43 | 47 | 48

14. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness and swelling at the injection site. Any = incidence of a particular symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) follow-up period after booster vaccination
Population: Analysis was performed on the Total Vaccinated cohort, which included all subjects with documented administration of Boostrix™ vaccine, any formulation, for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 55 | 59 | 62
Participants
  Any Pain | 50 | 55 | 54
  Any Redness | 23 | 23 | 21
  Any Swelling | 21 | 20 | 19

15. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms.
Description: Assessed solicited general symptoms were fatigue, gastrointestinal, headache and fever [defined as axillary temperature ≥ 37.5 degrees Celsius (°C)]. Any = incidence of a particular symptom regardless of intensity grade and relationship to vaccination.
Time Frame: During the 4-day (Days 0-3) follow-up period after booster vaccination
Population: as for outcome 14
Measure: Number; unit: subjects
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 59 | 62
subjects
  Any Fatigue | 17 | 20 | 22
  Any Gastrointestinal Symptoms | 10 | 9 | 13
  Any Headache | 13 | 19 | 13
  Any Fever | 1 | 1 | 1

16. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE is any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any unsolicited AE = any unsolicited AE regardless of intensity or relationship to vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up period after booster vaccination
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 55 | 60 | 62
Participants | 22 | 16 | 21

17. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject..
Time Frame: At Year 8.5
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 54 | 60 | 66
Participants | 0 | 0 | 0

18. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs).
Description: as for outcome 17
Time Frame: From Year 8.5 up to study end (one month post Year 10 booster vaccination)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Number analyzed (Participants) | 55 | 60 | 62
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs): Entire study period (From Year 8.5 to one month post Year 10) ; Unsolicited adverse events (AEs): During the 31 days (Day 0 - Day 30) post Year 10 booster vaccination; Solicited symptoms: During the 4 days (Day 0 - Day 3) post Year 10 booster vaccination.
Description: Total numbers of subjects at risk for SAEs are those at time points with highest numbers of subjects enrolled. For unsolicited and solicited AEs they correspond to the numbers of subjects with available results. Numbers at risk are the highest ones, at Year 8.5 for Boostrix-US Group, & Year 10 for the other groups.
Arm/Group | Boostrix-US Group | Boostrix-INV Group | Boostrix-REF Group
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/60 | 0/66
Other Adverse Events (participants affected / at risk) | 53/55 | 58/60 | 58/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Boostrix-US Group (N=55) | Boostrix-INV Group (N=60) | Boostrix-REF Group (N=62)
Nasopharyngitis (Infections and infestations) | 6 | 1 | 4 — Unsolicited AE reported among subjects receiving the Booster dose of vaccine administered at Year 10.
Headache (Nervous system disorders) | 5 | 1 | 3 — Unsolicited AE reported among subjects receiving the Booster dose of vaccine administered at Year 10.
Pain (General disorders) | 50 | 55/59 | 54 — Solicited local symptom assessed in and reported by subjects receiving the Booster dose of vaccine administered at Year 10.
Redness (General disorders) | 23 | 23/59 | 21 — Solicited local symptom assessed in and reported by subjects receiving the Booster dose of vaccine administered at Year 10.
Swelling (General disorders) | 21 | 20/59 | 19 — Solicited local symptom assessed in and reported by subjects receiving the Booster dose of vaccine administered at Year 10.
Fatigue (General disorders) | 17/54 | 20/59 | 22 — Solicited general symptom reported by subjects who received Year 10 booster vaccination and with available results.
Gastrointestinal symptoms (General disorders) | 10/54 | 9/59 | 13 — Solicited general symptom reported by subjects who received Year 10 booster vaccination and with available results.
Headache (General disorders) | 13/54 | 19/59 | 13 — Solicited general symptom reported by subjects who received Year 10 booster vaccination and with available results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.